CLINICAL TRIAL: NCT02890290
Title: Nutrition and Sarcopenia in Frail Elderly: a Randomized Controlled Trial of the Effects of Marine Protein Hydrolysates to Improve Physical Performance.
Brief Title: Effect Study of Marine Protein Hydrolysates to Prevent Loss of Muscle Mass and Physical Function in Frail Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molde University College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Nygard8362
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Sarcopenia
Keywords: Frail Elderly; Diet, Food, and Nutrition; physical function; marine protein hydrolysates; protein intake; seafood intake; ageing; old; nutrition; frail
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator): Marine protein hydrolysate pills (3000mg)
  Interventions: Dietary Supplement: Marine Protein hydrolysate
- Control (Placebo Comparator): Placebo pills (gum arabicum)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Marine Protein hydrolysate — The participants will take the supplement in form of tablets and will be instructed to take five tablets twice a day, preferably in relation to meals, however, not the dinner meal. Each tablet contains 300 mg of marine protein hydrolysates (Nx6.25). The tablets are produced by Flexipharma AS.
  Arms: Intervention
Dietary Supplement: Placebo — Placebo tablets will be made based on gum arabicum. The tablets are produced by Flexipharma AS.
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether a marine protein hydrolysate given as a supplement can prevent age related loss of muscle mass and loss of physical function in frail elderly. The study will recruit elderly living at home with help from municipal health care services, and a secondary goal of the study is to describe food habits, seafood intake and nutritional status in this group of patients.

Edit: the recruitment procedure was changed in august 2017, to include elderly without help from municipal health care services. Participants are now recruited trough media and organizations for elderly, and these changes in recruitment procedure was approved by the ethics committee august 2017.

DETAILED DESCRIPTION:
The overall objective in this project is to study how nutrition influences frailty and physical function in home-dwelling elderly.

The study will seek to answer the following hypotheses (RCT):

1. Sarcopenia as measures by SPPB, grip strength, antropometry and gait speed is significantly associated with nutritional status and intake of protein in frail elderly.
2. A supplement of 3000mg of marine peptides pr. day in 12 months in the intervention group will improve the score on SPPB and other sarcopenia-related outcomes like grip strength, antropometric measures or gait speed compared to the placebo group.

To supplement the results of the RCT, interviews will be performed with selected participants to answer the following question:

- How do frail elderly describe their own nutritional status and need of help from municipal health care service related to nutrition? The data collection will be made in the participants' home at baseline and after 6 and 12 months. The patients will complete the Short Physical Performance Test (SPPB), Grip Strength measurement and anthropometric measurements (weight, height, calf circumference and mid-arm circumference). Assessment of nutritional status will be made by Mini Nutritional Assessment (MNA). Seafood intake and protein intake will be assessed by a food frequency questionnaire based on previously used and validated questionnaires. Daily energy intake will be estimated by a 24-hour multiple pass recall of food intake. Health related quality of life will be assessed by the EQ-5D-5L questionnaire (EuroQol). In addition, the participants will be asked to take blood tests to be analyzed for vitamin D, nutritional and inflammation markers.

Sample size and statistical power calculation The main outcome of this study is physical performance, measured on a 12 point ordinal scale; the SPPB. In accordance to previous studies, a clinical meaningful change in score on this scale is 0,4 - 1,5 points. Based on mean values and SD from the mentioned study, power was computed with SPSS (IMB) Power Sample for t-test of independent samples. The criterion for significance (alpha) has been set at 0,050 and the test is 2-tailed. With a sample size of 39 in each of the two groups, the study will have a power of 80% to yield a statistically significant result. This computation assumes a difference between groups of 0.9 points. As the participants are frail and of old age, we expect a dropout/missing frequency of 20 %, thus we should have 50 participants in each group.

Statistical analyzes The null hypothesis is that there is no difference between intervention and control group, in change of physical performance across multiple test attempts. Linear mixed model will be used to detect differences in treatments across multiple test attempts. Linear mixed model and ordinal regression models will be used to explore the relationship between nutrition and physical performance at baseline.

In-depth interviews Interviews will provide a deeper understanding of potential results in the RCT. Fifteen to twenty participants will be selected to the interviews by purposeful recruitment, based on results from the RCT study. The interviews will be transcribed and analyzed using qualitative content analysis.

Ethical consideration This project was approved by the Regional Committee in Ethics in Medical Research in Mid- Norway. The investigators do not anticipate this project causing any harm or discomfort to the participants, and will make sure that our participants participate in the study voluntarily. Participants will be given both oral and written information about the study twice before they give their consent to participate. First, they will receive information from their home care nurse, and if they agree to receive a call or visit from the researcher, they will have the opportunity to ask questions before signing the written consent. Participants not receiving municipal health care services sign their consent at the first visit. Furthermore, they will be informed about the possibility to withdraw from the study without any consequences at any time.

The project will have considerable benefits for this patient group. Increased knowledge of the nutritional status and protein intake in the patient group may facilitate nutritional interventions to prevent loss of physical function, potentially leading to increased independence and delayed need of residential institution. Results from the RCT may be transferable to other patient conditions where muscle atrophy is expected, e.g. inactivity after injuries, bed rest after surgery, or in intensive care units.

ELIGIBILITY:
Inclusion Criteria:

* able and willing to give consent
* Must be able to swallow tablets

Exclusion Criteria:

* diabetes (recieve treatment)
* active cancer illness
* progressive muscle illness (e.g. multiple sclerosis ALS)
* kidney failure
* short life expectancy (<1år)
* allergies of fish protein.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 92 (Actual)
Dates: Start 2016-09; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) | 6 and 12 months
  physical test assessing balance, lower limb function and gait speed.

SECONDARY OUTCOMES:
Grip strength | 6 and 12 months
  Measured in kg with dynamometer
Gait speed | 6 and 12 months
  m/s calculated from 4 meter walking test in SPPB
Health related quality of life | 6 and 12 months
  as measured by EQ-5D-5L
Antropometric measures | 6 and 12 months
  see protocol

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Freiberger E, de Vreede P, Schoene D, Rydwik E, Mueller V, Frandin K, Hopman-Rock M. Performance-based physical function in older community-dwelling persons: a systematic review of instruments. Age Ageing. 2012 Nov;41(6):712-21. doi: 10.1093/ageing/afs099. Epub 2012 Aug 10. PMID 22885845
- [Background] Dodds RM, Syddall HE, Cooper R, Benzeval M, Deary IJ, Dennison EM, Der G, Gale CR, Inskip HM, Jagger C, Kirkwood TB, Lawlor DA, Robinson SM, Starr JM, Steptoe A, Tilling K, Kuh D, Cooper C, Sayer AA. Grip strength across the life course: normative data from twelve British studies. PLoS One. 2014 Dec 4;9(12):e113637. doi: 10.1371/journal.pone.0113637. eCollection 2014. PMID 25474696
- [Background] Kwon S, Perera S, Pahor M, Katula JA, King AC, Groessl EJ, Studenski SA. What is a meaningful change in physical performance? Findings from a clinical trial in older adults (the LIFE-P study). J Nutr Health Aging. 2009 Jun;13(6):538-44. doi: 10.1007/s12603-009-0104-z. PMID 19536422
- [Derived] Nygard LAK, Mundal I, Dahl L, Saltyte Benth J, Rokstad AMM. Nutrition and physical performance in older people-effects of marine protein hydrolysates to prevent decline in physical performance: a randomised controlled trial protocol. BMJ Open. 2018 Oct 8;8(10):e023845. doi: 10.1136/bmjopen-2018-023845. PMID 30297351